CLINICAL TRIAL: NCT00366756
Title: Evaluation of a Visual Acuity Testing Software for Children, VisionQuest 20/20
Brief Title: Evaluation of VisionQuest 20/20, a Visual Acuity Testing Software
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: M. Edward Wilson, Medcial University of South Carolina
Other Study IDs: SEI-06-001
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2010-12

CONDITIONS: Visual Acuity
Keywords: Vision; Visual Acuity

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study involves the use of VisionQuest 20/20 which is a new software program to test visual acuity in children. The purpose of this study is to compare the results of VisionQuest 20/20 to two other ways to measure visual acuity. The two other tests are a standard eye exam by an ophthalmologist and electronic visual acuity (EVA) testing, a computerized version of a standard eye test.

It is important to identify vision problems in children as early as possible. These problems include amblyopia ("lazy eye," or reduced vision due to lack of development in the visual area of the brain), strabismus (eyes are not aligned correctly due to eye muscle problems), and refractive errors (when you need glasses to see up close or far away). Early identification of the vision problems allows them to be treated earlier which makes it more likely that vision can be improved. VisionQuest 20/20 can be easily distributed to schools, and it is easy for the child and the vision screener to use. The test can be performed by volunteers instead of an ophthalmologist.

DETAILED DESCRIPTION:
Assessing visual acuity represents one of the most sensitive techniques for the detection of eye abnormalities in children. Vision disorders are the fourth most common disability in the USA and are the most prevalent handicapping condition in childhood. Ocular conditions, if undetected or untreated, can have substantial long-term implications for the quality of life of the child and the family and can place a burden on public health resources.

Important causes of visual impairment in children include amblyopia, strabismus and significant refractive error. Children with these conditions may benefit from early detection to allow treatment. Early detection and treatment is the key for successful management of children with visual disorders. If detected during childhood, treatment for amblyopia is effective and inexpensive. Although amblyopia is a treatable disorder if detected in childhood during the brain's "critical period" for vision development, every year the problem goes undetected and untreated in thousands of US children resulting in permanent visual disability for the individuals and hundreds of millions of dollars of annual economic loss to society. Furthermore, other less serious types of childhood vision problems, such as refractive errors, may contribute to academic underperformance if not identified during childhood. What ages, venues, and methodologies are best to perform vision screenings and when full eye examinations are indicated remains to be determined. , Nevertheless, nearly universal agreement exists among U.S. government agencies, health experts, educators, and charitable vision organizations that children should be screened for visual disorders, even if asymptomatic. To date, a combination of scientific, logistical, economic, and legislative shortcomings have prevented vision screening goals from being met for many U.S. children.

The ideal vision screening method should be accurate (sensitive and specific for clinically significant visual problems amenable to treatment), standardized, easy to administer and interpret with little training, cost effective, universally available to children, and capable of collecting data to ensure medical follow-up is received by those who need it as well as to collect epidemiological information and monitor the success of the program year after year. The Amblyopia Foundation of America (AFA) has conceptualized how automated computer software which assesses vision while a child "plays" a video game could potentially meet the requirements for an ideal vision screening system for children old enough to cooperate.

Young children are increasingly familiar with computers and videogames, oftentimes being more sophisticated in their use than their parents. Vision screening software is easy to distribute via CDs or the internet. Computers are readily available in virtually all schools and the cost of computer technology continues to decline even as performance improves. Computer software applications allow standardization of logic protocols for vision screenings and the videogame format allow for automated testing. Automated testing eliminates the need for large scale training and certification of vision screening proctors and instead can allow vision screenings to be performed by untrained lay volunteers or personnel already available in schools. Finally, since responses of children being tested are inputted directly into the computer, results may be printed instantaneously at the end of testing. Computer data may be warehoused locally or offsite via the internet to help coordinate medical follow-up for those children identified at risk, monitor the success of the program, and facilitate epidemiological analysis of vision disorders. Prototype VisionQuest 20/20 software currently performs standardized visual acuity assessments of each eye and stereopsis testing while a child "plays" a 2-3 minute video game.

A pilot study (O'Neil J.W., et al 2005 unpublished) suggested lay screeners using this an early version of this prototype vision screening software on laptop computers achieved similar positive and negative predictive value results to a certified ophthalmic technician using a professional grade M&S vision tester. Positive predictive values for clinically significant visual disorders were 54% for M&S and 52% for VisionQuest 20/20 respectively. Negative predictive values were identical at 97% for each screening method. VisionQuest 20/20 appears to have potential for use as a vision screener for schoolchildren and may allow more children to be reached than manual vision screening or other methods by relying on lay personnel already available in schools rather than certified vision screeners or eye professionals to perform screenings. Additional benefits include use of computers already available in schools with the potential to simplify vision screening logistics and reduce costs. Independent validity testing is essential before initiating large scale community vision screenings with this new vision screening software. The primary aim of the current study is to validate VisionQuest 20/20 screening software by assessing its ability to screen for threshold visual acuities as compared to an exact visual acuity obtained with the EVA tester using ETDRS optotypes. The secondary aim of the current study is to evaluate the ability of VisionQuest 20/20 software to detect the presence or absence of clinically significant vision disorders in children as compared to a professional eye examination by a pediatric ophthalmologist.

ELIGIBILITY:
Inclusion Criteria:

* 8-15 years of age
* healthy volunteers

Exclusion Criteria:

* significant developmental delays or motor skill impairments which would prevent children from independently operating a computer mouse
* psychiatric disorders and/or attention deficit disorder

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children ages 8-5 years with myopia.
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2006-07; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Standard Eye Test | 12 Months
  This study involves the use of VisionQuest 20/20 which is a new software program to test visual acuity in children. The purpose of this study is to compare the results of VisionQuest 20/20 to two other ways to measure visual acuity. The two other tests are a standard eye exam by an ophthalmologist and electronic visual acuity (EVA) testing, a computerized version of a standard eye test.

CONTACTS AND LOCATIONS:
Overall Officials: Marion E. Wilson, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Storm Eye Institute, Medical University of South Carolina, Charleston, South Carolina, United States